CLINICAL TRIAL: NCT04829851
Title: Personalised Nutrition for Healthy Living: The PROTEIN Project
Brief Title: The PROTEIN Project
Acronym: PROTEIN
Status: Completed | Type: Observational
Sponsor: University of Surrey (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Other Study IDs: PROTEIN
Record Dates: First submitted 2021-03-25; First posted 2021-04-02 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Overweight; Nutritional Deficiency; Poor Nutrition; Iron-deficiency
MeSH Terms: conditions — Overweight; Malnutrition; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Health Care Professionals: Registered health care professional, such as a General Practitioner/ Dietitian/ Nutritionist/ Registered Exercise Professional (REPs) etc. who sees clients for assistance with weight management and / or iron deficiency or diet quality.
  Interventions: Device: Expert Dashboard
- Adults who are Overweight: Adults (> 18 years) who are considered to be overweight (25 - 30 kg/m2) but are otherwise in good physical health and a regular android smart phone/ tablet user.
  Interventions: Device: PROTEIN Mobile App
- Adults with Iron Deficiency Anaemia: Adults (> 18 years) who have been diagnosed with Iron deficiency anaemia but are otherwise in good physical health and a regular android smart phone/ tablet user.
  Interventions: Device: PROTEIN Mobile App
- Adults with Low- Fruit/ Vegetable Intake: Adults ( > 18 years) with a low fruit and vegetable intake (2-3 portions/ d) but are otherwise in good physical health and a regular android smart phone/ tablet user.
  Interventions: Device: PROTEIN Mobile App

INTERVENTIONS:
Device: PROTEIN Mobile App — All recruited user groups will be expected to use the PROTEIN app. During this study the subjects will be asked to visit the lab followed by at least 4 weeks usage of the PROTEIN app and then a final lab visit.
  Groups: Adults who are Overweight; Adults with Iron Deficiency Anaemia; Adults with Low- Fruit/ Vegetable Intake
Device: Expert Dashboard — Health care professionals (HCP) will be contacted via email and will also be invited to either attend the lab or meet with the researchers utilizing Zoom/ Microsoft teams to discuss the usage of the expert dashboard within the PROTEIN application.
  Groups: Health Care Professionals

SUMMARY:
New advances in information computer technology and artificial intelligence (AI) offer the possibility to create a personalized tool and support system for healthy living and eating, and this is the principal objective of the PROTEIN Project (an EU-funded consortium; Horizon 2020). In order to obtain information on the acceptability, usability and its effectiveness at facilitating behaviour change of the application within the home and store. A pilot trial will be conducted in participants who are overweight (BMI 25-29.9 kg/m2) and a separate group of participants who consume a low quality diet (low in fruit and vegetable intake) and/or have a nutrition deficiency (specifically iron-deficiency anaemia).

During this study the subjects will be asked to attend the lab (or remotely due to covid restrictions) at the beginning of the study for baseline measurements and instructions on how to use / download the mobile application. Participants will have their anthropometrics measured (including height/ weight/ waist: hip circumference). The PROTEIN application will collect self-reported data from the user, which includes: user profile input, dietary and fluid intake, daily physical activity (such as step count), biochemistry, sleep and chewing (in- meal behaviour). Information on how users will interact with the app, which screens they use, how many log ons and how often data is inputted will also be collected. Throughout the trial, the participants will be contacted via the application or by the researchers to request feedback on their progress and to encourage reporting of any issues.

Health care professionals will also be recruited to test the expert dashboard of the PROTEIN app. Through this system they will be able to provide nutrition/ physical activity advice directly to their patients and input their relevant biochemical results (such as haemoglobin for anaemic patients).

DETAILED DESCRIPTION:
During this study the subjects will be asked to visit the lab followed between 4 and 16 weeks usage of the PROTEIN app and then a final lab visit.

In the event that COVID-19 restrictions continue and prevent, or restrict, face-to-face visits a completely remote study protocol will also be developed and used in place of the study below.

1. Advertising and Recruitment:

   i) General public: Prospective users will be recruited by the University of Surrey via social media (e.g. Facebook and Twitter), posters and flyers in the local area and emails sent to University staff and students. With the permission on the relevant group leaders,' overweight participants will be recruited via local commercial weight loss groups. With the permission of the practice managers recruitment via GP practices will also be undertaken, with practice registers screened by a member of practice staff and information/ invitation letters sent to those who meet the inclusion criteria (no details will be shared with the research team). Flyers will also be distributed to local relevant outpatient clinics, e.g. haematology and dietetic with the permission of the clinic managers.

   Participants will also be recruited through health care professionals (HCP) in the local area following identification of suitable HCPs (see below)

   ii) Health Care Professionals (HCPs):

   HCPs involved in supporting the dietary or activity goals of target clients will also be recruited to the HCP arm of the study. The project will be promoted through local (and, if remote, National) professional networks and professional body membership lists, newsletters and via relevant social media channels. HCPs will have the option to participate in a desk-based expert review of the application (without registering specific clients) with respect to its usability or to register one or more of their own clients on the app via the user dashboard to participate in the efficacy review. In the latter case suitable clients identified by the HCP will be required to also register with the trial. The HCP will be provided with flyers and invitation letters to allow them to make first contact with the client who will be asked to contact the research team to confirm their willingness to participate, ensuring no personal data is shared prior to consent being received.
2. Baseline measurements:

   i) Public, Face to face: Users will attend the lab and will then have their body composition measured (to include their height, weight, waist and hip circumference) by the researchers.

   ii) Public, Remote: An alternative remote protocol will utilise Zoom/ Microsoft teams video call. These will be arranged by the researchers with the participants to take them through self-completion of the baseline measures and procedures.

   iii) HCPs: HCPs will be contacted via email and will also be invited to either attend the lab or meet with the researchers utilizing Zoom/ Microsoft teams to discuss the usage of the expert dashboard.
3. PROTEIN app usage for public:

   Following this, the users will be requested to log the following details to set-up the PROTEIN system: contact details (name/ email/phone number), age, gender, height, weight, ethnicity, morbidity status (such as cardiovascular disease/ diabetes mellitus etc.), education/ socioeconomic status, smoking status, diet or drink habits (such as vegetarian/ vegan/ dairy-free etc.), and medication.

   Daily food and fluid intake will be collected via the PROTEIN app and will be self-reported by the user/ participant.

   Users will be asked to log all dietary and fluid intake for 7 days per week (to include the weekend) into the home PROTEIN application suite.

   Users will either use their respective smartwatches/activity trackers or manually input the relevant data into the home PROTEIN application suite. In the former case, physical activity and sleep data will be collected in daily summaries as provided by Google Fit (or a suitable alternative, such as Garmin, FitBit, Polar, Apple watch etc.).

   Smart watches may be provided free of charge for a subset of users (subject to trial resources) and there may also be an opportunity for participants to use their own existing smartwatches. In the latter case, users will be requested to manually log daily activity data, for 7 days per week.

   Users will be monitored by the PROTEIN artificial intelligence (AI) system for deviations from their suggested plan and for any meal or activity swaps requested to check for adherence/ compliance to the recommendations suggested by the PROTEIN AI system.

   A subset of users who are also registered with OCADO will receive food shopping recommendations (in the form of a shopping list) tailored to their nutritional requirements and targets; budget will also be taken into account. Participants will be asked to indicate all food products that they swapped/ bought and for whom they bought them within the PROTEIN application suite. This will be conducted in partnership with OCADO.
4. After at least 4 weeks of usage, data will be collected regarding the user and HCP experience via an online questionnaire through the PROTEIN app or sent usability questionnaires via email by the researchers.
5. Follow-up measures:

   i) Public, Face to face: Users will attend the lab after at least 4 weeks of usage and will then have their body composition remeasured (to include their height, weight, waist and hip circumference) by the researchers. They will also be asked to provide feedback on the usability of the application by completing two questionnaires on the 1) usability of the application and 2) suitability for general public use.

   ii) Public, Remote: An alternative remote protocol will utilise Zoom/ Microsoft teams video call. These will be arranged by the researchers with the participants to take them through self-completion of the follow-up measures following at least 4 weeks of usage. Participants will be asked to provide feedback via two online questionnaires on the 1) usability of the application and 2) suitability for general public use.

   iii) HCPs: HCPs will be contacted via email and will also be invited to either attend the lab or meet with the researchers utilizing Zoom/ Microsoft teams to discuss their feedback following usage of the expert dashboard for at least 4 weeks. They will be asked to provide feedback via two questionnaires on the 1) usability of the application and 2) suitability for usage by health care professionals.

   A subset of participants (from all groups), representing both those who have engaged or not with the app, will also be contacted by the researchers after their trial period has ended and invited to take part in additional qualitative measures, such as focus group interviews to provide more feedback on their experience of the PROTEIN app.

ELIGIBILITY:
Inclusion Criteria:

Overweight group:

* ≥ 18 years of age
* BMI: 25 - 30 kg/m2
* In good physical health
* Not a regular user of another nutrition support application (such as MyFitnessPal)
* Able to provide written informed consent
* Android Smart Phone/ Tablet user

Individuals with poor quality diet

1. deficiencies:

   * ≥ 18 years of age
   * Diagnosed iron deficiency
   * In good physical health
   * Not a regular user of another nutrition support application (such as MyFitnessPal)
   * Able to provide written informed consent
   * Android Smart Phone/ Tablet user Individuals with poor quality diet
2. low fruit and vegetable intake:

   * ≥ 18 years of age
   * Low fruit and vegetable intakes (< 2-3 portions/ day)
   * In good physical health
   * Not a regular user of another nutrition support application (such as MyFitnessPal)
   * Able to provide written informed consent
   * Android Smart Phone/ Tablet user

Health care professionals

* Registered health care professional; General Practitioner/ Dietitian/ Nutritionist/ Registered Exercise Professionals (REPs) etc who sees clients for assistance with weight management and/ or iron deficiency or diet quality.
* Willing to trial a new nutrition support application with their patients
* Android Smart Phone/ Tablet user

Exclusion Criteria:

Overweight group:

* Those who have been diagnosed with cardiovascular disease, type 1 diabetes mellitus or type 2 diabetes mellitus.
* Currently receiving treatment for long term medical conditions
* Clinically significant haematological abnormalities or an active malignancy
* Regular exercisers (more than 150 minutes of moderate exercise per week or > 75 minutes of high intensity exercise)
* People who are unable to exercise for medical reasons or for whom exercise is otherwise contra-indicated by a health professional
* People with disordered eating (such as anorexia nervosa etc.)
* Those who are not be able to provide written consent.
* Those who are unable to read/write sufficiently to provide consent and complete study materials

Individuals with deficiencies and poor-quality diet:

* Those who have been diagnosed with cardiovascular disease, type 1 diabetes mellitus or type 2 diabetes mellitus.
* Currently receiving treatment for long term medical conditions.
* Clinically significant haematological abnormalities or an active malignancy
* Regular exercisers (more than 150 minutes of moderate exercise per week or > 75 minutes of high intensity exercise)
* People who are unable to exercise for medical reasons or for whom exercise is otherwise contra-indicated by a health professional
* People with disordered eating (such as anorexia nervosa etc.)
* Those who are not be able to provide written consent.
* Those who are unable to read/write sufficiently to provide consent and complete study materials

Health Care Professionals:

* Not affiliated/ registered health care professional
* Do not have any clients/ patients that fall into one of the groups above (overweight, iron deficiency or low fruit/ vegetable consumption).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General public within the local area (Surrey, UK)
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of the PROTEIN mobile application's ability to facilitate a lifestyle change | At least 4 weeks
  Users will be requested to set up the application on their smartphone / tablet, following this the users will be provided with a suggested plan through the artificial intelligence (AI) system. Users will be asked to log all dietary and fluid intake for 7 days per week into the PROTEIN application suite. Therefore, the primary outcome measure will be the adherence/ compliance to the recommendations suggested by the PROTEIN AI system following up to 4 weeks of usage of the mobile application.

SECONDARY OUTCOMES:
Shopping acceptability within the application | At least 4 weeks
  A subset of users who are also registered with OCADO will receive food shopping recommendations (in the form of a shopping list) tailored to their nutritional requirements and targets: budget will also be taken into account. Users will be asked to indicate the acceptability of this function within the mobile application after at least 4 weeks of usage.
Efficacy of the PROTEIN application to monitor within-meal chewing | At least 4 weeks
  Within-meal behaviours will be analysed through the application on at least 4 separate occasions during their 4-week usage of the application. The users will be asked to record themselves eating a meal within the PROTEIN application, which will calculate their chew count. Therefore, the efficacy of the system will be ealuated for within-meal chewing behaviours by all users.
User Satisfaction with the PROTEIN Application | At least 4 weeks
  A subset of participants (from all groups), representing both those who have engaged or not with the app, will be contacted by the researchers after their trial period has ended and invited to take part in additional qualitative measures, such as focus group interviews to provide more user satisfaction feedback on their experience of the PROTEIN application.
Suitability and usability review of the PROTEIN application for Health Care Professionals | At least 4 weeks
  Health care professionals (HCP) will be involved in supporting the dietary or activity goals of target clients recruited. HCPs will have the option to participate in a desk-based expert review of the application (without registering specific clients) with respect to its usability or to register one or more of their own clients on the app via the user dashboard to participate in the efficacy review. They will be asked to provide feedback via two questionnaires on the 1) usability of the application and 2) suitability for usage by health care professionals.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Surrey, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No